CLINICAL TRIAL: NCT06337227
Title: Potential Role of Sirtuins As Epigenetic Biomarkers for the Clinical Management of the Patient with Atherosclerosis or Calcific Aortic Stenosis
Brief Title: Potential Role of Sirtuins As Epigenetic Biomarkers of the Patient with Atherosclerosis or Calcific Aortic Stenosis
Status: Recruiting | Type: Observational
Sponsor: IRCCS SYNLAB SDN (Other)
Collaborators: Federico II University (Other)
Responsible Party: Sponsor
Other Study IDs: 2/22
Record Dates: First submitted 2024-03-22; First posted 2024-03-29 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Atherosclerosis and Calcific Aortic Stenosis with and Without Diabetes
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- atherosclerosis and calcific aortic stenosis with diabetes patients
  Interventions: Diagnostic Test: lncRNA signature analyses
- atherosclerosis and calcific aortic stenosis without diabetes patients
  Interventions: Diagnostic Test: lncRNA signature analyses
- Patients without atherosclerosis undergoing surgical procedure for endocarditis
  Interventions: Diagnostic Test: lncRNA signature analyses

INTERVENTIONS:
Diagnostic Test: lncRNA signature analyses — Specific validation experiments will be performed by Real-Time PCR (C-reactive protein), Western Blot, flow cytometry and microscopy

SUMMARY:
The project aims to shed light on the role of Sirtuins, enzymes belonging to the third class of histone deacetylases (class III) involved in epigenetic modifications (deacetylation), focusing mainly on Sirtuin 6 (SIRT6), as a regulator of atherosclerosis and severe aortic valve stenosis through molecular-based and epigenetic studies in human VSMC cells.

ELIGIBILITY:
Inclusion Criteria:

* Patients with atherosclerosis or calcific aortic stenosis with and without diabetes older than 18 years of either sex;
* Patients without atherosclerosis undergoing surgical procedure for endocarditis;
* Patients who will have signed informed consent

Exclusion Criteria:

* Patients for whom biological material cannot be recovered for study purposes;
* Patients who refuse to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study plans to recruit 100 patients admitted to AOU Federico II Cardiac Surgery in Naples subject to surgical procedure with atherosclerosis and calcific aortic stenosis with and without diabetes over a 36-month period. Patients without atherosclerosis or aortic valve stenosis will be considered as a control population and where possible included in a statistical design paired for age and sex with the study population
Sampling Method: Probability Sample
Enrollment: 3 (Estimated)
Dates: Start 2023-10-19 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
To evaluate by analysis of data obtained from NGS techniques whether and which proteins belonging to the Sirtuin family may be deregulated in patients with atherosclerosis or calcific aortic stenosis | 36 months

SECONDARY OUTCOMES:
To evaluate the experimental results achieved in the clinical-diagnostic context | 36 months

CONTACTS AND LOCATIONS:
Locations (1):
- Irccs Synlab Sdn, Naples, Italy

IPD SHARING:
Plan to Share IPD: No